CLINICAL TRIAL: NCT02876640
Title: Phase Ib 9cUAB30 in Early Stage Breast Cancer to Evaluate Biologic Effect
Brief Title: Retinoid 9cUAB30 in Producing a Biologic Effect in Patients With Early Stage Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate Accrual Rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2016-01293; NCI-2016-01293 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00033; UW16063 (Other: University of Wisconsin Carbone Cancer Center - University Hospital); UWI2015-05-01 (Other: DCP); N01CN00033 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2024-05-22 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Breast Ductal Carcinoma In Situ; Early Stage Breast Carcinoma; Invasive Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Specimen Handling; UAB 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (retinoid 9cUAB30) (Experimental): Patients receive retinoid 9cUAB30 PO QD for 14 to 28 days. Patients then undergo tumor resection surgery. Patients undergo blood and urine sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Retinoid 9cUAB30; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Retinoid 9cUAB30 — Given PO
  Other Names: (9Z)-UAB-30; 9cUAB30; UAB-30
Procedure: Therapeutic Conventional Surgery — Undergo tumor resection surgery

SUMMARY:
This phase 1b trial studies the biologic effect of 9cUAB30 on early stage breast cancer. 9cUAB30 is a retinoid X receptor (RXR)-selective retinoid that acts in a tissue selective manner with the goal of minimizing side effects, a necessary feature of agents under development for cancer prevention.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare molecular analysis of pre- and post-treatment tissue samples of breast cancers of patients treated with 14-28 days of oral retinoid X receptor (RXR)-selective retinoid 9cUAB30 (9 cUAB30) will demonstrate significantly reduced proliferation.

SECONDARY OBJECTIVES:

I. Determine if 14-28 days of oral RXR-selective 9c-UAB30 treatment increases apoptotic index, as measured by cleaved caspase 3 assay.

II. Examine the differences in gene expression from baseline to post-exposure breast cancer samples using a custom gene panel from Nanostring Technologies.

III. To examine if the maximum concentration (Cmax) and safety of 9cUAB30 in the first 5 participants is affected by reducing the number of capsules at the 240 mg dose level.

IV. To examine the Cmax of all participants at baseline and on the day of surgery.

V. Determine if treatment with 2-4 weeks of 9cUAB30 prior to surgery will increase gene expression of type I immune cells in the tumor immune environment of all participants except the first 5.

VI. Assess the overall safety of 9cUAB30 in comparison with known retinoid toxicity.

EXPLORATORY OBJECTIVE:

I. Determine if treatment with 2-4 weeks of 9cUAB30 prior to surgery will increase activated type I dendritic cells in peripheral blood.

OUTLINE:

Patients receive retinoid 9cUAB30 orally (PO) once daily (QD) for 14 to 28 days. Patients then undergo tumor resection surgery. Patients undergo blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed up at 7 days and 4-5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female only. The sample size of males affected by breast cancer is limited, hence we will not be able to collect significant data for analysis of the effect of study drug on breast cancer in males
* Age >= 18 years. Because no dosing or adverse event data is currently available on the use of 9cUAB30 in participants <18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 or Karnofsky >= 70%
* Invasive breast cancer diagnosed by needle core biopsy between 0.5 cm and 5 cm in size based on imaging, that is estrogen receptor positive (ER+) or estrogen receptor negative (ER-), Her2neu positive or negative OR ductal carcinoma in situ (DCIS) of the breast diagnosed by core needle biopsy and at least 1.0 cm in size based on imaging. Grade 3 ER+ DCIS will be allowed as well as ER- DCIS of any grade. For DCIS-only lesions, the imaging abnormality corresponding to the cancer must be at least 1.0 cm in size (i.e. calcifications, distortion or mass on mammogram, or mass or non-mass enhancement on magnetic resonance imaging [MRI])
* White blood cells (WBC) >= 3000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin > 10 g/dL
* Bilirubin =< upper limit of institutional normal
* Aspartate aminotransferase (AST) =< upper limit of institutional normal
* Creatinine =< upper limit of institutional normal
* Triglycerides =< 1.5 x upper limit of normal (ULN)
* Cholesterol =< 1.5 x ULN
* Participants must agree to discontinue all supplements containing vitamin A while taking study medication and for thirty days after the last dose of study medication.
* Have not been treated with chemotherapy, or biological therapy in the last 5 years. We do not know if the previous treatment will have an effect on the tissues to be examined.
* Have not used tamoxifen, raloxifene, or other antiestrogen compounds within 6 months of study entry. If used within 5 years of study entry, total duration of use must be less than 6 months
* Have not used exogenous hormone replacement therapy or hormonal contraception in the year prior to diagnosis. The use of non-systemic estrogen (such as vaginal estrogen use) is allowed
* The effects of 9cUAB30 on the developing human fetus are unknown. Since retinoids are known to be teratogenic, to avoid any complications due to unintentional pregnancies only postmenopausal women and some premenopausal women (as outlined below) will be eligible; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

  * Women will be considered postmenopausal if one of the following is met:

    * Prior bilateral oophorectomy
    * 60 years of age or older
    * Age less than 60 years; amenorrheic for 12 or more months; and follicle stimulating hormone (FSH) in the postmenopausal range
  * Premenopausal women without childbearing potential are eligible to participate if one of the following criteria is met:

    * Prior hysterectomy
    * Prior fallopian tubal ligation (cut, tied, or sealed)
    * Prior placement of permanent intratubal contraceptive devices (e.g. Essure)
    * Partner with prior vasectomy and willing to use barrier method (e.g. condoms)
* Participants must have the ability to understand, and the willingness to sign, a written informed consent document

Exclusion Criteria:

* Participant taking medications that might interact with 9cUAB30
* Participant who has started or increased dosage of lipid-lowering agents in the last 30 days of enrollment
* Participant receiving any other investigational agents within 30-days of enrollment nor during study participation with the exception of 18F-FFNP investigational imaging agent
* Participant with a history of allergic reactions attributed to compounds of similar chemical or biologic composition of retinoids
* Participant with an uncontrolled intercurrent illness including, but not limited to;

  * Ongoing or active infection,
  * Symptomatic congestive heart failure,
  * Unstable angina pectoris,
  * Cardiac arrhythmia,
  * A persistent grade 3 hypertension

    * For grade 1, grade 2, and non-persistent grade 3 hypertension, repeat blood pressure reading after 5 minutes. If the average reading of the two measurements is grade 3 (systolic BP >=160 mm Hg or diastolic BP >=100 mm Hg) the patient is not eligible. If the average reading of the two measurements is less than or equal to grade 2, then the participant is eligible. If the average of the 2 readings is grade 1 or grade 2 hypertension, document the appropriate level hypertension on the baseline symptom form.
  * Psychiatric illness/social situations that will limit compliance with study requirements
* Participant who is breastfeeding or planning to breastfeed for a month post last dose of study agent
* Participant known to be human immunodeficiency virus (HIV)-positive, as we do not know the effects of study drug on suppression of the immune system.
* Participant with a history of a second cancer diagnosis or reoccurrence < 2 years from study entry with the exception of a history of squamous or basal cell carcinoma of the skin < 2 years from study entry will not be excluded from this study. This is to eliminate the residual effects of any previous treatments for those cancers
* Participant with history of ipsilateral breast radiation
* Participant's core biopsy slides suggest that later re-sectioning will not contain sufficient tumor to allow for an adequate evaluation of Ki67 and caspase 3 assays, at a minimum

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Krontiras, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Northwestern University, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Thomas PS, Patel AB, Lee JJ, Liu DD, Hernandez M, Muzzio M, Contreras A, Sepeda V, Mays C, Weber D, Vornik LA, Khan SA, Dimond E, Heckman-Stoddard BM, Perloff M, Brown PH. Phase I Dose Escalation Study of Topical Bexarotene in Women at High Risk for Breast Cancer. Cancer Prev Res (Phila). 2023 Jan 4;16(1):47-55. doi: 10.1158/1940-6207.CAPR-22-0210. PMID 36228112

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Retinoid 9cUAB30)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-64 years | 14
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.97 (6.95)
Respirations [Mean (Standard Deviation); unit: breaths per minute] | 15.74 (1.65)
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 3
  Post-menopausal | 24
Time from Diagnosis to study Entry [Mean (Standard Deviation); unit: days] | 32.85 (19.14)
Breast Cancer Location [Count of Participants; unit: Participants]
  Left Breast | 13
  Right Breast | 14
Breast Cancer Biology [Count of Participants; unit: Participants]
  Invasive Lobular Carcinoma | 4
  Invasive Ductal Carcinoma | 20
  Invasive Mammary Carcinoma | 3
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Negative | 3
  Positive | 24
HER2 IHC Result [Count of Participants; unit: Participants] — HER2 IHC reporting came from the initial diagnostic biopsy. This is a clinical datapoint with no variation of severity. IHC 0 or 1 indicate HER2-negative. IHC 2 is equivocal. IHC 3 indicates HER2- positive. Population: 3 of the cancers were estrogen receptor negative
  Participants
    number analyzed (Participants) | 22
    0 | 14
    1+ | 5
    2+ | 2
    3+ | 1
Estrogen Receptor Score [Mean (Standard Deviation); unit: percentage] — This is a results obtained from the clinical pathology report from the participants' initial biopsy. The method of assessment is based on clinical pathological analysis.
  percentage | 85.96 (31)
HER2 FISH [Count of Participants; unit: Participants] — This is a result obtained from the clinical pathology report from the participants initial biopsy. The method of assessment is based on clinical pathological analysis.
  Participants
    Equivocal | 1
    No result/not done not amplified | 26

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Ki-67 Expression in Breast Epithelial Cells of Patients Treated With 9cUAB30
Description: Ki-67 was analyzed using immunohistochemistry. Absolute change was measured in looking at the baseline in comparison to that at the end of treatment.
Time Frame: Baseline up to 28 days (post-exposure)
Population: One participant's sample did not have any tumor tissue to be analyzed
Measure: Mean (Standard Deviation); unit: Percent of cells
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 26
Percent of cells | 0.2 (3.7)

2. Secondary Outcome: Change in Apoptosis in Breast Epithelial Cells of Patients Treated With 9cUAB30
Description: Will be assessed by caspase 3 assays and immunohistochemistry. Change between the treated and matched controls will be summarized with descriptive statistics. Difference in apoptosis will be compared between treatment and matched "control" group using a one-tailed paired t-test or Wilcoxon signed-rank test, as appropriate, at a significance level of 0.05.
Time Frame: Baseline up to 28 days (post-exposure)
Population: One participant's sample did not have any tumor tissue to analyze
Measure: Mean (Standard Deviation); unit: percent of cells
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 26
percent of cells | 0.62 (2.75)

3. Secondary Outcome: Change in Gene Expression of Breast Cancer Samples Using a Custom Gene Panel From Nanostring Technologies
Description: Change in gene expression will be summarized with descriptive statistics.
Time Frame: Baseline up to 28 days (post-exposure)
Measure: Mean (Full Range); unit: % of protein
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 27
% of protein
  Up regulated IL6 expression | 9.49 [4.85 to 18.60]
  Down regulated CDKN2A expression | 0.34 [0.254 to 0.617]

4. Secondary Outcome: Change in Maximum Concentration (Cmax)
Description: Will be tested by a one-sided one-sample student t-test.
Time Frame: Pre-dose, 5 minutes, and 2 hours post-dose
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 27
ng/mL | 990.7 (312.9)

5. Secondary Outcome: Incidence of Observed Adverse Events
Description: Will be graded according to Common Terminology Criteria for Adverse Events version 4.0. Will be compared to know retinoid toxicity. These will be described in descriptive statistics and analyzed.
Time Frame: Up to 28 days
Measure: Number; unit: number of adverse events
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 27
number of adverse events | 128

6. Secondary Outcome: Change in Activated Type I Dendritic Cells in Peripheral Blood
Time Frame: Baseline up to 28 days (post-exposure)
Population: 19 patients had matched pre and post samples
Measure: Mean (Standard Deviation); unit: percent of cells
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 19
percent of cells
  type 1 CD40+mDCs | 0.12 (0.22)
  CD86+ mDCs | 1.0 (8.71)
  type 1 CD86+ macrophages | -0.15 (0.26)
  HLADR+ pDCs | -6.42 (12.11)
  CD33+CD11b+HLA DR+ CD40+ cells | 0.26 (0.78)

7. Secondary Outcome: Determine if Treatment With 2-4 Weeks of 9cUAB30 Prior to Surgery Will Increase Gene Expression of Type I Immune Cells in the Tumor Immune Environment of All Participants
Time Frame: Baseline up to 28 days (post-exposure)
Population: Data was not collected
Arm/Group | Treatment (Retinoid 9cUAB30)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Treatment (Retinoid 9cUAB30)
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 26/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Retinoid 9cUAB30) (N=27)
constipation (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 4
dry mouth (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 2
fatigue (General disorders) | 10
malaise (General disorders) | 2
venous injury (Injury, poisoning and procedural complications) | 2
cholesterol high ldl (Investigations) | 5
Cholesterol non-hdl high (Investigations) | 6
white blood cell decreased (Investigations) | 2
hypertriglyceridemia (Metabolism and nutrition disorders) | 2
back pain (Musculoskeletal and connective tissue disorders) | 2
headache (Nervous system disorders) | 8
dry skin (Skin and subcutaneous tissue disorders) | 2
pruritis (Skin and subcutaneous tissue disorders) | 3
rash acneiform (Skin and subcutaneous tissue disorders) | 4
rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
hypertension (Vascular disorders) | 14
Cholesterol high (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT02876640/Prot_SAP_000.pdf